CLINICAL TRIAL: NCT04761965
Title: Clinical Study of the Sensitivity and Specificity of the Quantitative Assessment of Bone Marrow Cellularity by MRI in Comparison With Trepanobiopsies in Patients With Diseases of the Hematopoietic System
Brief Title: Quantitative MRI of Bone Marrow Fat Fraction in Patients With Trepanobiopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCPHOI-2019-06
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Aplastic Anemia; Aplastic Anemia Idiopathic
Keywords: Quantitative MRI; trepanobiopsy; Aplastic Anemia Idiopathic; children
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone marrow cellularity by mDixon-quant — if trepanobiopsy was performed during the diagnosis, then comparison with MRI Bone marrow cellularity by mDixon-quant

SUMMARY:
The study is aimed to find correlation between the assessment of cellularity according to trepanobiopsy data and the results of measuring MRI parameters.

DETAILED DESCRIPTION:
The ratio of fat to water in the bone marrow depends on the cellularity of the bone marrow. In addition to the water/fat ratio in bone marrow there are also other parameters for quantitative MRI assessment. These include the apparent diffusion coefficient (ACD), the T1 relaxation time, mapping of the macromolecular proton fraction. The undoubted advantage of MRI is its non-invasiveness and the ability to assess any localization of the bone marrow.

MRI may become a new non-invasive method for assessing the cellularity of the bone marrow in children with oncohematological diseases.

ELIGIBILITY:
Inclusion Criteria:

presence of indications for performing trepanobiopsy:

1. aplastic anemia
2. chronic myeloproliferative disease
3. reactive changes in hematopoiesis

Exclusion Criteria:

1. Refusal to sign an informed consent to participate in a clinical trial
2. Presence of contraindications for MRI examination
3. Extremely serious condition of the patient at the time of inclusion in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
correlation between Bone marrow cellularity by mDixon-quant and trepanobiopsy. | Before the start of treatment
  Determination of bone marrow cellularity before starting therapy for the underlying disease. Cellularity according to trepanobiopsy data is the ratio of stromal and hematopoietic cells to fat cells in the bone marrow. Cellularity according to MRI - the ratio of water and fat in the bone marrow using the mDixom Quant.

SECONDARY OUTCOMES:
T1 maping | Before the start of treatment
  T1 mapping (ms) is a magnetic resonance imaging technique used to calculate the T1 time
apparent diffusion coefficient | Before the start of treatment
  value of apparent diffusion coefficient in mm2/s
Percentage of the macromolecular proton fraction (MPF) | Before the start of treatment
  Percentage of the macromolecular proton fraction (MPF)
Percentage of the bone marrow fat fraction | Before the start of treatment
  Percentage of the bone marrow fat fraction (FF) by spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow, Samory-Mashela,1, Russia

IPD SHARING:
Plan to Share IPD: No